CLINICAL TRIAL: NCT00827489
Title: Ascending Single Dose Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of HTC-867 Administered Orally to Healthy Subjects
Brief Title: Study Evaluating HTC-867 in Healthy Young and Elderly Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3253A1-1000
Record Dates: First submitted 2009-01-21; First posted 2009-01-22 (Estimated); Last update posted 2009-09-02 (Estimated); Status verified 2009-09

CONDITIONS: Healthy Subjects
Keywords: schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- HTC-867 (Experimental)
  Interventions: Drug: HTC-867
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: HTC-867
  Arms: HTC-867
Other: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and tolerability of ascending single oral doses of HTC-867 in healthy young and elderly subjects. This study will also evaluate the way the drug enters and leaves the blood and tissues over time and how the drug acts on and in the body in a fasted and fed state.

ELIGIBILITY:
Inclusion:

1. Men or women of nonchildbearing potential (WONCBP) aged 18 to 50 years or 65 or greater inclusive at screening.

   WONCBP may be included if they are either surgically sterile (hysterectomy and/or oophorectomy) or postmenopausal for ≥1 year (with follicle-stimulating hormone [FSH] ≥38 mIU/mL) and must have a negative pregnancy test result within 48 hours before administration of study drug.

   Women who are surgically sterile must provide documentation of the procedure by an operative report or by ultrasound scan.

   Sexually active men must agree to use a medically acceptable form of contraception during the study and continue it for 12 weeks after study drug administration.
2. Healthy as determined by the investigator on the basis of screening evaluations.
3. The elderly subjects must be generally healthy, but may be enrolled with a stable, chronic illness if it is well controlled and does not interfere with the primary objective of the study. Subjects may be included with clinically important deviations from normal limits in medical history, physical examination findings, vital sign measurements, 12-lead electrocardiograms (ECGs), or clinical laboratory test results that are associated with stable, chronic, and well-controlled medical conditions, so long as those deviations do not meet the stated specific criteria for exclusion

Exclusion:

1. Presence or history of any disorder that may prevent the successful completion of the study.
2. History of cardiac disorders (other than hypertension) including but not limited to valvular disease, congestive heart failure, angina pectoris, myocardial infarction, or arrhythmia.
3. History of vertigo.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Safety as measured by the number of adverse events and serious adverse events. Tolerability as measured by occurrence of dose limiting toxicities. | 5 months

SECONDARY OUTCOMES:
Pharmacokinetic and pharmacodynamic parameters. | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Overland Park, Kansas, United States